CLINICAL TRIAL: NCT00939744
Title: Study of the Effect of Eicosanoids on Contractile Activity of Pregnant Human Myometrium in Pathological Situation.
Acronym: EAU2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, MD, PhD, Dr, Université de Sherbrooke
Other Study IDs: 09-040
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Obstetric Labor Complications; Prolonged Pregnancy
Keywords: contractile activity; eicosanoids; pregnant women; obstetrics complications
MeSH Terms: conditions — Obstetric Labor Complications; Pregnancy, Prolonged

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — uterus biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EAU2: Women who will have a c-section at the CHUS

SUMMARY:
Recent studies show that EET and 20-HETE have important biological effects, particularly in the vascular system. The investigators studied the effect of eicosanoids on the gravid rat uterus. The results suggest that 20-HETE had an tocolytics effect on gravid uterus. In the previous study, we demonstrated that the enzymes of the pathway of EET were present in human uterine tissues. Moreover, the addition of an inhibitor of degradation of EET had an tocolytic effect on the human myometrium, as the exogenous addition of 8.9, 14,15-EET and 20-HETE.

Objectives:

Primary objective: To compare the balance of different metabolic pathways of arachidonic acid (AA) of the pregnant human myometrium in pathological situations (preterm labor, uterine atony, prolonged pregnancy).

Specific objectives: i) To study the effect of derived from the AA on in vitro contractile activity of normal and pathological uterine tissues, and ii) detect and quantify the different sub-products of metabolism of AA in the uterine tissues (myometrium, fetal membranes and placenta).

The management of uterine contraction is in the heart of modern obstetrics year, yet the progress made in other specialties, based on the study of smooth muscle have not yet been transposed in obstetrics. A better understanding of systems for regulating the contraction is important in terms of 1) new physiological knowledge, but it could also be the source of 2) modification of strategies to take care of premature delivery (new Tocolytic), or 3) improving the efficiency of uterine muscle during delivery or 4) for treatment of patients with prolonged pregnancy.

DETAILED DESCRIPTION:
It is a clinical study with a slope fundamental aims to examine the metabolic pathways of AA of human myometrium and their functional roles according to their clinical profile divided into three contractile pathological situations - threat of premature delivery, dynamic dystocia, prolonged pregnancy - and two groups of patients at term: a group before work and group work.

The sampling method. After birth, a biopsy will be perform from the lower segment of the uterus. After caesarean sections of membrane and placenta are collected.

The substances studied during isometric tension tests are part of the three degradation pathways of the AA.

1. new eicosanoids in cumulative dose (8,9-EET, 11,12-EET, 14,15-EET, 20-HETE), and in combination
2. enzyme inhibitors of the eicosanoids pathway (AUDA, MS-PPOH, DDMS), and the COX and LOX pathways (indomethacin), alone or in combination.

ELIGIBILITY:
Inclusion Criteria:

* all women who will have a c-section

Exclusion Criteria:

* induction of labor,
* child with malformation,
* birth weight less than 2500 grams or greater than 4500g

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women who will have a c-section at the CHUS
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2009-05; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
effect of eicosanoids on contractile activity of myometrium of pregnant women with pathological situations | during c-section

SECONDARY OUTCOMES:
effect of enzymatic inhibitors on contractile activity of myometrium from pregnant women with pathological situations | during c-section
detection of enzymes from the different pathways | after c-section
quantification of eicosanoids in different tissues | after c-section

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Sherbrooke; Rousseau Éric, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier de l'Université de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Corriveau S, Pasquier JC, Blouin S, Bellabarba D, Rousseau E. Chronic levothyroxine and acute T3 treatments enhance the amplitude and time course of uterine contractions in human. Am J Physiol Endocrinol Metab. 2013 Mar 1;304(5):E478-85. doi: 10.1152/ajpendo.00346.2012. Epub 2012 Dec 18. PMID 23249699